CLINICAL TRIAL: NCT06189365
Title: Amplatzer Amulet China Post Market Study (PMS)
Status: Terminated | Type: Observational
Why Stopped: This study was terminated due to the shift in Sponsor's business strategy.
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10491; CRD_1028 (Other: Abbott)
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-Valvular Atrial Fibrillation
Keywords: Non-Valvular Atrial Fibrillation; NVAF; Amplatzer Amulet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Amplatzer Amulet LAA occluder: Subject will receive the Left Atrial Appendage (LAA) closure procedure with Amplatzer Amulet LAA occluder.
  Interventions: Device: Left Atrial Appendage (LAA) closure procedure with Amplatzer Amulet LAA occluder

INTERVENTIONS:
Device: Left Atrial Appendage (LAA) closure procedure with Amplatzer Amulet LAA occluder — Subject will receive the Left Atrial Appendage (LAA) closure procedure with Amplatzer Amulet LAA occluder.

SUMMARY:
The purpose of this study is to prospectively evaluate the safety and effectiveness of the Amplatzer Amulet LAA occluder in a Chinese patient population indicated for use of this device.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained heart rhythm disorder. During AF, chaotic electrical activity results in rapid, uncoordinated, and insufficient contractions of the atrial chambers. Stagnation of blood flow in the left atrium (LA) can lead to hypercoagulability. The left atrial appendage (LAA), given its location and complex shape is often the primary site of stasis and thus increases the risk for thrombus formation. Approximately 90% of all thrombi in patients with non-valvular AF (NVAF) forming in the LA originate in the LAA.

Patients with NVAF are at an increased risk of systemic embolism and stoke due to the potential for clot forming in the LAA. OAC is the recommended first-line therapy for NVAF at increased risk of stroke, however, many patients have relative or absolute contraindications to taking OACs. LAAO offers a non-pharmacological option for stroke risk reduction in these patients unable to take OAC.

The Amulet occluder is Abbott's second-generation LAA occlusion device. It received CE Mark in 2013, and FDA approval in August 2021. Observational studies performed in multiple geographies show that the Amulet occluder can be safely implanted with good procedural outcomes and reduce the risk of stroke as compared to a predicted rate without the need for anticoagulation in most patients. This led to the National Medical Products Administration (NMPA) approval of the Amulet occluder in 2020.

The purpose of this study is to prospectively evaluate the safety and effectiveness of the Amplatzer Amulet LAA occluder in a Chinese patient population indicated for use of this device.

ELIGIBILITY:
Inclusion Criteria:

1. Documented non-valvular atrial fibrillation and contraindicated for long-term oral anticoagulation, or in those who are taking oral warfarin but still develop stroke or relevant events
2. Meets the current device indications and per physician discretion for Amulet implant
3. Able to provide written Informed Consent prior to any study related procedures
4. 18 years of age or older at the time of enrolment

Exclusion Criteria:

1. With the presence of intracardiac thrombus
2. With active endocarditis or other infections producing bacteremia
3. Patients whose low risk of stroke (CHA2DS2-VASC score is 0 or 1) or bleeding (HAS-BLED score < 3)
4. Where placement of the device would interfere with any intracardiac or intravascular structures
5. Has a life expectancy of less than 2 years due to any condition
6. Currently participating or planning on participating during the follow up period of this study in a clinical study that includes an active treatment arm or a concurrent clinical study which may confound the results of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This clinical investigation will enroll subjects of all genders from the Chinese nationality general population ≥18 years old. Patients must meet all general eligibility criteria and provide written informed consent prior to sites conducting any investigation-specific procedures not considered standard of care.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of major adverse events | 7 days
  The primary short-term safety endpoint is the occurrence of one or more of the following major adverse events within 7 days after the procedure: all-cause mortality, procedure or device-related complications requiring open cardiac surgery or major endovascular intervention, ischemic or hemorrhagic stroke, or systemic embolism.
Occurrence of device embolization,device erosion,clinically significant device interference with surrounding structure, device thrombus, device fracture, device related infections(endocarditis and pericarditis), device breakage, or device related allergy | 2 years
  The primary long-term safety endpoint is the occurrence of device embolization, device erosion, clinically significant device interference with surrounding structure, device thrombus, device fracture, device related infections (endocarditis and pericarditis), device breakage, or device related allergy through 2 years.
Composite of ischemic stroke or systemic embolism | 2 years
  The primary effectiveness endpoint is a composite of ischemic stroke or systemic embolism through 2 years.

OTHER OUTCOMES:
Rate of ischemic stroke or systemic embolism | 5 years
  Rate of ischemic stroke or systemic embolism through 5 years post-implant
Composite of damage to blood vessel or organ or damage to adjacent organs at implant, device dislodgement, device fracture, device erosion, or pericardial tamponade | 5 years
  Composite of damage to blood vessel or organ or damage to adjacent organs at implant, device dislodgement, device fracture, device erosion, or pericardial tamponade through 5 years post-procedure
Rate of device success | During implant procedure, approximately 30 to 60 minutes
  Rate of device success - defined as device deployed and implanted in correct position
Rate of device closure | 3 months
  Rate of device closure - defined as residual jet around the device of ≤ 5mm, based on the 3 month transesophageal echocardiogram (TEE) defined by Doppler flow
Percentage of subjects taking OAC or antiplatelet drugs | 5 years
  Percentage of subjects taking OAC or antiplatelet drugs through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhihui ZHANG, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (5):
- China (5):
  - University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Zhuzhou Central South University, Zhuzhou, Hunan
  - Xianyang Hospital Of Yan'an University, Xianyang, Shaanxi

IPD SHARING:
Plan to Share IPD: No